CLINICAL TRIAL: NCT06565013
Title: Impact of Increased Patient Engagement Associated With Cabotegravir (CAB) + Rilpivirine (RPV) Long-acting (LA) Administered Every Two Months on Virologically Suppressed People Living With HIV Who Are Practicing Chemsex
Brief Title: Chemsex Health Evaluation With Extended Release System for HIV Treatment
Acronym: CHEERS
Status: Not yet recruiting | Type: Observational
Sponsor: Clinique Médicale L'Actuel (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ACT001
Record Dates: First submitted 2024-07-17; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: HIV
Keywords: Chemsex; Global health; Linkage to care; Switch; Vulnerable population; Long-acting; Patient Reported Outcomes
MeSH Terms: conditions — Chemsex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CHEERS main: Switch from daily oral ART to Cabenuva, administered IM every two months.
  * Cabotegravir: 200mg/ml, 3ml per dose
  * Rilpivirine: 300mg/ml, 3ml per dose
  Interventions: Drug: Cabenuva 600/900; Other: Self administered questionnaires; Other: Semi-directed interview

INTERVENTIONS:
Drug: Cabenuva 600/900 — Participants will switch to Cabenuva at baseline. The visit schedule, the product administration and the clinical follow-up will be done according to standard of care.
Other: Self administered questionnaires — Questionnaires on treatment satisfaction (HIVTSQs), quality of life (WHOQoL-HIV-BREF) and drug use assessment (DEBA-D) will be administered at baseline, M5 and M11
Other: Semi-directed interview — At baseline and M11, participants will conduct a semi-directed interview about the perception of their HIV treatment and the global care they receive as a person living with HIV who is practicing chemsex.

SUMMARY:
CHEERS is an observational cohort for people living with HIV who are actively practicing chemsex and who are switching to CAB + RPV LA after being virologically suppressed on a stable oral ART regimen. This study aim to assess the impact of increased patient engagement associated with this LA regimen on linkage to psychosocial care and on global health outcomes, such as quality of life, substance use, treatment satisfaction and virological control.

Eligible participants will need to be currently out of care for psychosocial counselling and will need to express the wish to switch to CAB + RPV LA. The participants will be followed in this study for 11 months from their first LA administration, according to the schedule of injections. In addition to standard of care procedures, such as blood draw and physical exam, patient reported outcome questionnaires will be administered at certain visits and a semi-directed interview will be conducted at the beginning and at the end of the study. CAB + RPV LA will be used in line with the Canadian monography.

ELIGIBILITY:
Inclusion Criteria

1. Man, trans-woman or gender diverse person who was assigned male at birth and is over 18 y.o.
2. Actively practices chemsex, as assessed by self-reported use of substances (methamphetamine, GHB/GBL, ketamine and mephedrone) as a mean of prolonging sexual relations, intensifying sexual pleasure and/or exploring one's sexual subjectivity at least once in the last month prior to screening*.
3. Living with HIV-1 and virologically suppressed (plasma HIV RNA < 50 c/ml) on stable oral ART regimen for at least one month prior to screening.
4. Not currently receiving psychosocial support, either on site or outside of the clinic, as evaluated by an absence of self- reported psychosocial consultation in the last 3 months prior to screening.
5. Participant is capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
6. Participant is able to locally source Cabenuva, as this product is not provided in the context of this study.

   * If a patient only tried it once and it occurred in the last month prior to screening, we will consider that they meet the inclusion criteria, although we will focus on enrolling patients with a documented history of regular substance use, as pre-identified by chart review.

Exclusion Criteria

1. History or presence of allergy, resistance or intolerance to Cabotegravir or Rilpivirine, or drugs of their class.
2. Exposure to an experimental drug or experimental vaccine within 30 days prior to first dose of study treatment.
3. Alanine aminotransferase (ALT) 5 times the upper limit of normal (ULN); or ALT 3xULN and bilirubin 1.5xULN (with >35% direct bilirubin).
4. Participant has estimated creatine clearance <30mL/min per 1.73 m2
5. Any concomitant condition or medication prohibited by local prescribing information.
6. Any condition judged by the investigator that may interfere with the study or the patient's well being if they were being enrolled.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults living with HIV on daily oral ART who are actively practicing chemsex and who are not currently involved in a psychosocial follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of psychosocial linkage | From baseline through month 11
  This study aims to demonstrate the impact of a switch to Cabenuva on patient engagement by measuring linkage to psychosocial care. The investigators will assess the proportion of participants who complete at least one psychosocial visit during the study.

SECONDARY OUTCOMES:
Change in the HIV Treatment Satisfaction Questionnaire (HIVTSQ) score | Baseline, month 5 and month 11
  This study aims to assess the reported treatment satisfaction before and after a switch to Cabenuva by measuring the change in HIVTSQs scores. The sacle is from 0 to 6.A higher score is associated with a higher satisfaction.
Change in discourse on treatment and care satisfaction | Baseline and month 11
  This study aims to assess the reported treatment satisfaction before and after the switch to Cabenuva by measuring the change in perception of HIV treatment and care, as assessed by a semi-directed interview. Thematic content analysis (TCA) will be used to identify changes. The investigators will evaluate the change for people who initiated a psychosocial follow-up and for those who didn't.
Change in the WHO Quality of life HIV questionnaire (brief version) | Baseline, month 5 and month 11
  This study aim to assess the perceived quality of life before and after a switch to Cabenuva, as measured by change in WHOQoL-HIV-BREF (quality of life questionnaire) score throughout the study. the scale score is from 4-20.A higher score is associated with a higher quality of life.
Frequency and severity of drug use | Baseline, month 5 and month 11
  This study aim to assess the frequency and severity of drug use before and after switch to Cabenuva, as measured by the change in DEBA-D (drug use assessment questionnaire) score throughout the study. The scale score is from 0-15. A higher score is associated with a more frequent and severe use of drugs.
Frequency of detectable viremia | 24 months prior to baseline as well as from baseline through month 11
  This study aim to assess the change in frequency of detectable viremia before and after the switch to Cabenuva in a vulnerable population.
Attendance rate to clinical visits | Up to 24 months prior to baseline and from baseline through month 11
  This study aim to characterize the span of patient engagement as assessed by the change in attendance rate to clinical visits before and after switch to Cabenuva.
Frequency rate of psychosocial visits | Up to 24 months prior to baseline and from baseline through month 11
  This study aim to characterize the span of patient engagement as assessed by change in frequency of psychosocial visits before and after switch to Cabenuva (only applicable to participants who had previously disengaged from psychosocial care and who initiated a psychosocial follow-up in the context of this study).
  For each participant, we will compare the frequency rate of psychological visits they attended during the 24 months before screening to the frequency of visits they attended during the 11-month period from baseline (Day 1) to Month 11. We anticipate three possible outcomes:
  The frequency rate of psychological visits increased, The frequency rate of psychological visits decreased, or The frequency rate of psychological visits stayed the same.
Number of psychosocial visits | From baseline through month 11
  This study aim to characterize the span of patient engagement as assessed by the number of psychosocial visits per participant who engage in care.
Discontinuation rate | From baseline through month 11
  This study aim to characterize the span of patient engagement as assessed by the discontinuation rate to both clinical and psychosocial visits.
Proportion of visits done outside window | From baseline through month 11
  This study aim to characterize the span of patient engagement as assessed by the proportion of clinical visits done outside the visit window.
Frequency of AEs (safety) | From baseline through month 11
  This study aim to assess the safety of Cabenuva in this population by evaluating the frequency of serious AE or drug related AEs, including site injection reactions.
Proportion of viral failure | From baseline until the date of confirmed viral failure, assessed up to month 11
  This study aim to assess the maintenance of viral suppression by evaluating the proportion of viral failure at the end of the study.
Incidence of viral resistance development | From baseline until the date of confirmed viral failure, assessed up to month 11
  For participants experiencing viral failure, this study aims to assess whether there is a development of drug resistance specifically to cabotegravir and rilpivirine.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Szabo, MD, PhD, Principal Investigator — Clinique Médicale L'Actuel
Locations (1):
- Clinique Médicale l'Actuel, Montreal, Quebec, Canada